CLINICAL TRIAL: NCT00174018
Title: Validity and Reliability in Measuring the Subacromial Space by Using Ultrasound
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261700931
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-12-07 (Estimated); Status verified 1993-08

CONDITIONS: Shoulder Impingement
Keywords: subacrominal space
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
To investigate validity and reliability in measuring the subacrominal space by using ultrasound

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects age range 19-35 years

Exclusion Criteria:

* With any pain in the upper extremities and back

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 1993-09

CONTACTS AND LOCATIONS:
Overall Officials: Hsing-Kuo Wang, PhD, Study Director — School and Graduate institute of Physical Therapy, National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, NTU, Taiwan, Taipei, Taiwan